CLINICAL TRIAL: NCT07026760
Title: Effects of Trans-spinal Magnetic Stimulation on Cortical Excitability in Healthy Individuals
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Kátia Monte-Silva, Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 58678222.8.0000.5208
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Healthy Individuals
Keywords: Trans-spinal magnetic stimulation; Cortical Excitability

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Trans-spinal magnetic stimulation (1 Hz + 90% MT) (Active Comparator)
  Interventions: Device: Trans-spinal magnetic stimulation (90% MT + 1 Hz)
- Trans-spinal magnetic stimulation (1 Hz + 100% MT) (Active Comparator)
  Interventions: Device: Trans-spinal magnetic stimulation (100% MT + 1 Hz)
- Trans-spinal magnetic stimulation (1 Hz + 110% MT) (Active Comparator)
  Interventions: Device: Trans-spinal magnetic stimulation (110% MT + 1 Hz)
- Trans-spinal magnetic stimulation (10 Hz + 90% MT) (Active Comparator)
  Interventions: Device: Trans-spinal magnetic stimulation (90% + 10 Hz)
- Trans-spinal magnetic stimulation (10 Hz + 100% MT) (Active Comparator)
  Interventions: Device: Trans-spinal magnetic stimulation (100% MT + 10 Hz)
- Trans-spinal magnetic stimulation (10 Hz + 110% MT) (Active Comparator)
  Interventions: Device: Trans-spinal magnetic stimulation (110% MT + 10 Hz)
- Trans-spinal magnetic stimulation (25 Hz + 90% MT) (Active Comparator)
  Interventions: Device: Trans-spinal magnetic stimulation (90% MT + 25 Hz)
- Trans-spinal magnetic stimulation (25 Hz + 100% MT) (Active Comparator)
  Interventions: Device: Trans-spinal magnetic stimulation (100% MT + 25 Hz)
- Trans-spinal magnetic stimulation (25 Hz + 110% MT) (Active Comparator)
  Interventions: Device: Trans-spinal magnetic stimulation (110% MT + 25 Hz)

INTERVENTIONS:
Device: Trans-spinal magnetic stimulation (90% MT + 1 Hz) — Low frequency stimulation (1 Hz) at 90% of resting motor threshold intensity, delivering a total of 2400 pulses.
  Arms: Trans-spinal magnetic stimulation (1 Hz + 90% MT)
Device: Trans-spinal magnetic stimulation (100% MT + 1 Hz) — Low frequency stimulation (1 Hz) at 100% of resting motor threshold intensity, delivering a total of 2400 pulses.
  Arms: Trans-spinal magnetic stimulation (1 Hz + 100% MT)
Device: Trans-spinal magnetic stimulation (110% MT + 1 Hz) — Low frequency stimulation (1 Hz) at 110% of resting motor threshold intensity, delivering a total of 2400 pulses.
  Arms: Trans-spinal magnetic stimulation (1 Hz + 110% MT)
Device: Trans-spinal magnetic stimulation (90% + 10 Hz) — High frequency stimulation (10 Hz) at 90% of resting motor threshold intensity, delivering a total of 2400 pulses.
  Arms: Trans-spinal magnetic stimulation (10 Hz + 90% MT)
Device: Trans-spinal magnetic stimulation (100% MT + 10 Hz) — High frequency stimulation (10 Hz) at 100% of resting motor threshold intensity, delivering a total of 2400 pulses.
  Arms: Trans-spinal magnetic stimulation (10 Hz + 100% MT)
Device: Trans-spinal magnetic stimulation (110% MT + 10 Hz) — High frequency stimulation (10 Hz) at 110% of resting motor threshold intensity, delivering a total of 2400 pulses.
  Arms: Trans-spinal magnetic stimulation (10 Hz + 110% MT)
Device: Trans-spinal magnetic stimulation (90% MT + 25 Hz) — High frequency stimulation (25 Hz) at 90% of resting motor threshold intensity, delivering a total of 2400 pulses.
  Arms: Trans-spinal magnetic stimulation (25 Hz + 90% MT)
Device: Trans-spinal magnetic stimulation (100% MT + 25 Hz) — High frequency stimulation (25 Hz) at 100% of resting motor threshold intensity, delivering a total of 2400 pulses.
  Arms: Trans-spinal magnetic stimulation (25 Hz + 100% MT)
Device: Trans-spinal magnetic stimulation (110% MT + 25 Hz) — High frequency stimulation (25 Hz) at 110% of resting motor threshold intensity, delivering a total of 2400 pulses.
  Arms: Trans-spinal magnetic stimulation (25 Hz + 110% MT)

SUMMARY:
This study investigates the immediate effects of different parameters (frequency and intensity) of trans-spinal magnetic stimulation (TsMS) on cortical excitability in healthy individuals. Using a randomized, double-blind crossover design, the research aims to identify optimal stimulation protocols for modulating neural activity. Outcomes include measurements of motor-evoked potentials (MEP), intracortical inhibition (ICI), and facilitation (ICF). Findings may enhance non-invasive therapeutic strategies for neurological disorders.

DETAILED DESCRIPTION:
This clinical trial comprises one arm: it evaluates trans-spinal magnetic stimulation (TsMS) applied at the C7 vertebral level, testing three frequencies (1 Hz, 10 Hz, and 25 Hz) and three intensities (90%, 100%, and 110% of the resting motor threshold) across sequential phases.

Methods: The study is a crossover, double-blind trial in which healthy adults (aged 18-40 years) undergo pre- and post-intervention assessments of cortical excitability (MEP, ICI, and ICF). Statistical analyses will be performed using ANOVA or Friedman tests (SPSS v.26).

The results will clarify whether the neuromodulatory effects of the stimulation are parameter-dependent and will guide future rehabilitation protocols for neurological conditions.

The research was approved by the Ethics Committee of the Federal University of Pernambuco (Resolution 466/12). All data will be stored securely for the next five years.

ELIGIBILITY:
Healthy adults aged 18-40 years, of both sexes; right-handed (confirmed via the Edinburgh Handedness Inventory); and for women, consistent use of contraceptive medication to mitigate hormonal influences on nervous system excitability.

Exclusion Criteria:

Pregnancy; history of seizures or epilepsy; metallic implants in the head, spine, face, or heart; diagnosed neurological or musculoskeletal conditions that could interfere with assessments or interventions; or use of substances that alter nervous system excitability.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Cortical excitability | Baseline (T0), immediately post-stimulation (T1), and at 15 (T2) and 30 minutes (T3) after stimulation.
  Cortical excitability will be assessed using motor-evoked potentials (MEPs) elicited by single-pulse transcranial magnetic stimulation (TMS) over the primary motor cortex (M1), specifically targeting the cortical representation of the first dorsal interosseous (FDI) muscle. The stimulation hotspot will be defined as the scalp location that elicits the largest and most consistent MEP amplitude at the lowest stimulation intensity. Single-pulse TMS will be delivered at 100% of the resting motor threshold (RMT). Paired-pulse TMS protocols will be used to evaluate intracortical inhibition (ICI) and intracortical facilitation (ICF), using a subthreshold conditioning stimulus set at 80% of RMT and a suprathreshold test stimulus set at 120% of RMT, with interstimulus intervals of 3 ms for ICI and 10 ms for ICF. MEP amplitudes will be recorded from the FDI muscle using bipolar surface electromyography (EMG). Signals will be digitized at 20,000 Hz (bandpass 5-10,000 Hz) for offlin

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No